CLINICAL TRIAL: NCT01251887
Title: Dietary Linoleic Acid Regulation of Omega-3 HUFA Metabolism: Satiety and Body Composition Among Overweight Female Subjects
Brief Title: Dietary Essential Fatty Acid Regulation of Omega-3 HUFA Metabolism; Satiety and Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 110028; 11-AA-0028
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2018-07-25

CONDITIONS: Weight Gain; Healthy Subjects; Obesity; Women
Keywords: Lipids; Obesity; Omega-3 Fatty Acids; Overweight
MeSH Terms: conditions — Weight Gain; Obesity; Overweight | interventions — Linoleic Acid; Docosahexaenoic Acids; Eicosapentaenoic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet A: Low omega-3 (n-3) + High linoleic acid (LA) (Experimental): Study diet containing 8 % energy (en%) linoleic acid (LA), 0.4 % energy (en%) arachidonic acid (AA), 0.05 % omega-3 highly unsaturated fatty acids (HUFA) for 12 weeks
  Interventions: Dietary Supplement: Linoleic Acid; Dietary Supplement: Docosahexaenoic Acid; Dietary Supplement: Eicosapentaenoic Acid
- Diet B: Low omega-3 (n-3) + Low linoleic acid (LA) (Experimental): Study diet containing 1 % energy (en%) linoleic acid (LA), 0.4 % energy (en%) arachidonic acid (AA), 0.05 % omega-3 highly unsaturated fatty acids highly unsaturated fatty acids (HUFA) for 12 weeks
  Interventions: Dietary Supplement: Linoleic Acid; Dietary Supplement: Docosahexaenoic Acid; Dietary Supplement: Eicosapentaenoic Acid
- Diet C: High omega-3 (n-3) + Low linoleic acid (LA) (Experimental): Study diet containing 1 % energy (en%) linoleic acid (LA), 0.4 % energy (en%) arachidonic acid (AA), 0.81 % omega-3 (n-3) HUFA for 12 weeks
  Interventions: Dietary Supplement: Linoleic Acid; Dietary Supplement: Docosahexaenoic Acid; Dietary Supplement: Eicosapentaenoic Acid

INTERVENTIONS:
Dietary Supplement: Linoleic Acid
Dietary Supplement: Docosahexaenoic Acid
Dietary Supplement: Eicosapentaenoic Acid

SUMMARY:
Background:

- Rates of obesity have increased dramatically in recent decades, and researchers are investigating how changes in diets and physical activity have contributed to this increase. To understand how weight might be controlled, it is important to learn what kinds of dietary changes can affect hunger and might lower body weight. Essential fatty acids, for instance, are an important part of a healthy diet, but researchers have not yet determined the ideal amount of essential fatty acids that people should eat. By studying how different diets affect body chemistry and hormone levels in women who are overweight or obese, researchers hope to be able to determine better diets or treatments to help people reach and maintain an optimum healthy weight.

Objectives:

- To examine how certain fats in the diet affect body metabolism, hormones, and weight regulation.

Eligibility:

- Healthy women between 18 and 50 years of age who are overweight or obese (body mass index between 25 and 35).

Design:

* This study has an initial screening visit and three phases. All participants will be involved in the first two phases of the study, and some participants will be involved in the third phase.
* Participants will be screened with a physical examination and medical history, in addition to blood and urine tests and questionnaires about eating habits and other diet factors.
* Phase 1: Participants will have three visits to the National Institutes of Health over a 4-week period. At the visits, participants will have blood and urine tests, complete questionnaires, and have other tests including brain and body imaging studies. Participants will then be assigned to one of three study diets.
* Phase 2: Participants will have a 12-week diet phase, with all foods supplied by the study researchers. Participants will keep a daily log of food and beverage intake, and will have three testing sessions with procedures similar to those performed in Phase 1.
* Phase 3: Participants assigned to a particular study diet (one-third of all participants) will be given the option of continuing the diet for an additional 36 weeks (9 months), with food consumption, monitoring, and testing procedures similar to those performed in Phase 2....

DETAILED DESCRIPTION:
Objective

To evaluate the effects of lowering the dietary nutrient linoleic acid (LA) as a controlled variable on: 1) tissue accretion of omega-6 and omega-3 highly unsaturated fatty acids (HUFA); 2) bioactive endocannabinoids derived from the omega-6 HUFA arachidonic acid (AA); 3) insulin sensitivity; 4) satiety and hunger; and 5) body composition. Modifications in dietary LA will be offset with reciprocal changes in the nutrient oleic acid (OA) to maintain equivalency of calories and nutrients.

Study Population

Up to 180 overweight, but otherwise healthy pre-menopausal women volunteers (aged 18 through 50) with body mass index (BMI) between 25 and 35 kg/m(2), will be enrolled.

With the anticipated dropout rates described in Section 7.4, we anticipate that 84 of these subjects will be randomized to study diets, and 64 subjects will complete the 12 week diet phase.

Three Group Comparative Analysis

A total of 84 subjects will be randomized to one of 3 healthy and nutritionally complete diets that differ only in the fatty acid composition of added visible oils. All foods will be provided through the NIH metabolic kitchen, with subjects visiting the kitchen daily Monday through Friday to obtain foods. Each Friday, subjects will carry home foods packed for their weekend meals. Baseline testing battery will include: 1) blood composition of omega-6 and omega-3 HUFA; 2) endocannabinoid, eicosanoid, and docosanoid derivatives of omega-6 and omega-3 HUFA; 3) insulin function assessment; 4) body composition assessment; 4) functional satiety assessment; and 5) self-reported measures of satiety, hunger and affective states. The full baseline testing battery will be repeated after 84 days of randomized treatment. An abbreviated testing battery will be performed after 28 and 56 days of randomized treatment.

A subset of participants will undergo additional inpatient testing in the 24-hour metabolic chamber as described in Section 3.3.2. The remaining subjects will remain ambulatory throughout the study. Participants will be advised to continue their usual medical care and medications throughout the study.

36-Week Continuation (Gradient Dose Replacement) Sub Study

At completion of the 84 day (12 week) study, participants in the low LA group (Group B) will have the option of continuing their study diets for another 252 days (36 weeks). During the continuation phase, the abbreviated testing battery will be completed after 6, 12, 18, 24 and 30 weeks, and the full testing battery will be repeated after 36 weeks.

Outcome Measures

A Primary Dependent Variables

The primary outcomes will be the proportion of omega-6 HUFA in total HUFA (%omega-6 in HUFA) and two endocannabinoids derived from omega-6 AA, 2-Arachidonoylglycerol (2-AG) and N-Arachidonoylethanolamine (Anandamide or AEA).

Secondary Dependent Variables

Secondary outcome measures will include blood concentrations of the omega-6 HUFA Arachidonic Acid (AA); the omega-3 HUFA Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA); the rates of change in %omega-6 in HUFA, AA, EPA, DHA, 2-AG and AEA over time; adipose and muscle tissue fatty acid composition; endocrine hormones; gene expression profiles; psychometrics; functional satiety; 24-hr energy metabolism and substrate utilization; and body composition, as follows: Omega-6 and omega-3 HUFA and total fat content will be measured in adipose and muscle tissue biopsies. Other endocannabinoid, eicosanoid and docosanoid derivatives of omega-6 and omega-3 HUFA will be measured in plasma via mass spectrometry.

Psychometric outcomes will include self-reported measures of satiety and affective states. Functional satiety will be assessed via buffet-style food array testing. Body composition outcomes will include DEXA, 3T MRI, anthropometric measurements and bioelectrical impedance. Genotyping will also be performed to assess for interactions between selected gene variants and effects of the intervention.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be overweight, but otherwise healthy, pre-menopausal ambulatory volunteers aged 18 to 50.

To be eligible for this research study, participants must:

* Be between 18 and 50 years of age.
* Have regular menstrual cycles.
* Be willing to use an effective method of birth control such as hormonal contraception, intrauterine device, barrier methods combined with spermicide, or surgical sterilization.
* Have a body mass index of 25 to 35 kg/m(2).
* Be otherwise healthy as determined by history, medical examination and laboratory tests.
* Be able to come to the NIH Clinical Center every weekday for 3 months.
* Be able to understand the consent form, and provide informed written consent.

EXCLUSION CRITERIA:

Participants are not eligible for this research study if they:

* Have been pregnant or have breast fed within the last 2 years.
* Work, or have an immediate family member who works, with a study investigator. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Are HIV positive.
* Have any current, unstable medical conditions including respiratory insufficiency requiring oxygen therapy; cardiac ischemia; cardiac or hepatic failure; or acute neurological illness as assessed by history and physical exam.
* Have evidence of diseases that may influence metabolism (e.g. overt diabetes mellitus, thyroid disease, cancer)
* Have any current or past history of eating disorders such as binge eating or anorexia nervosa.
* Have had weight loss (bariatric) surgery.
* Have gained or lost more than 3% of your current weight in the past 3 months.
* Exercise strenuously, like running, swimming, or basketball, 4 or more times per week.
* Are planning to begin a strenuous exercise program in the next 4 months.
* Take supplements that contain omega-6 or omega-3 fatty acids (e.g. fish, cod liver, borage, evening primrose oils)
* Have significant dietary limitations (e.g. multiple food allergies/intolerances, vegan diet) or special dietary requirements that are difficult to accommodate with study diets
* Have significant claustrophobia that would preclude study tests.
* Have a history of alcohol or substance abuse or dependence in the past 5 years.
* Drink more than 2 alcoholic beverages per day, on average, or 6 drinks per sitting in the past year. Participants may drink up to one alcoholic beverage per day during the study.
* Used marijuana, amphetamines, cocaine, or heroin even once over the last year. Participants may not use marijuana, amphetamines, cocaine, or heroin during the study.
* Have smoked 2 or more cigarettes per week, on average, over the past year.
* Participants may not use tobacco products during the study.
* Eat fish 3 or more times per week on average.
* Have a known bleeding disorder.
* Take medications or supplements that may interfere with this study by altering energy metabolism, nutrient absorption, or food intake. Regular use of the following compounds warrants exclusion: medications for the management of diabetes (Type 1 or 2), typical and atypical antipsychotics, thyroid medications, glucocorticoids, orlistat, decongestants, anti-histamines, and medications for cardiac conditions (e.g. beta blockers), attention disorders (e.g. amphetamine derivatives), blood lipid disorders (e.g. statins, fibrates), and hypertension (e.g. thiazide diuretics), as well as certain anti-depressants (e.g. tricyclics), and supplements that impact energy metabolism, such as ephedrine.
* Regularly take an anticoagulant medication, such as warfarin or aspirin.
* Have a pacemaker, brain stimulator, or other implanted electrical device, permanent eyeliner, metallic prosthesis (including metal pins and rods, heart valves, and cochlear implants) that would preclude MRI scans.
* Are currently participating in any other clinical research studies that include blood draws or other procedures.
* Have a serum follicle-stimulating hormone (FSH) level greater than 20 units per liter

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2010-11-12; Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Ramsden, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cota D. The role of the endocannabinoid system in the regulation of hypothalamic-pituitary-adrenal axis activity. J Neuroendocrinol. 2008 May;20 Suppl 1:35-8. doi: 10.1111/j.1365-2826.2008.01673.x. PMID 18426497
- [Background] Pagotto U, Marsicano G, Cota D, Lutz B, Pasquali R. The emerging role of the endocannabinoid system in endocrine regulation and energy balance. Endocr Rev. 2006 Feb;27(1):73-100. doi: 10.1210/er.2005-0009. Epub 2005 Nov 23. PMID 16306385
- [Background] Szmitko PE, Verma S. The endocannabinoid system and cardiometabolic risk. Atherosclerosis. 2008 Aug;199(2):248-56. doi: 10.1016/j.atherosclerosis.2008.03.011. Epub 2008 Mar 20. PMID 18440538

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 85 subjects were consented to protocol. 19 of the 85 subjects were screen failures and one subject cancelled prior to start of study due to scheduling conflict.
Period: Overall Study
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Started | 18 | 29 | 18
Completed | 17 | 26 | 16
Not Completed | 1 | 3 | 2
Not completed — Scheduling conflict | 1 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA) | Total
Number analyzed (Participants) | 18 | 29 | 18 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 29 | 18 | 65
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 29 | 18 | 65
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 3 | 8
  Not Hispanic or Latino | 17 | 24 | 15 | 56
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 11 | 8 | 27
  White | 8 | 13 | 4 | 25
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of n-6 HUFA in Total HUFA (%n-6 in HUFA)
Description: Tissue accretion of omega-6 (n-6) highly unsaturated fatty acids (HUFA) in fasting plasma as percent of total HUFA.
Time Frame: Baseline
Population: The analyses included only those participants who completed at least 4 weeks of the diet phase with fasting blood samples available
Measure: Least Squares Mean (Standard Error); unit: Percentage of total HUFA
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total HUFA | 80.0 (1.2) | 81.3 (0.9) | 80.5 (1.1)

2. Primary Outcome: Proportion of n-6 HUFA in Total HUFA (%n-6 in HUFA)
Description: Tissue accretion of omega-6 (n-6) highly unsaturated fatty acids (HUFA) in fasting plasma as percent of total HUFA.
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total HUFA
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total HUFA | 80 (1.1) | 80.7 (0.9) | 70.6 (1.1)

3. Primary Outcome: Proportion of n-6 HUFA in Total HUFA (%n-6 in HUFA)
Description: Tissue accretion of omega-6 (n-6) highly unsaturated fatty acids (HUFA) in fasting plasma as percent of total HUFA.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total HUFA
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total HUFA | 79.7 (1.2) | 80.6 (0.9) | 70.8 (1.1)

4. Primary Outcome: Proportion of n-6 HUFA in Total HUFA (%n-6 in HUFA)
Description: Tissue accretion of omega-6 (n-6) highly unsaturated fatty acids (HUFA) in fasting plasma as percent of total HUFA.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total HUFA
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total HUFA | 80.6 (1.1) | 81 (0.9) | 72.9 (1.1)

5. Secondary Outcome: Proportion of n-6 HUFA Arachidonic Acid (AA)
Description: Tissue accretion of Arachidonic Acid (AA or 20:4n6), an omega-6 (n-6) highly unsaturated fatty acid, as measured in fasting plasma as a percent of total fatty acids.
Time Frame: Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 6.42 (0.3) | 6.51 (0.22) | 7.12 (0.29)

6. Secondary Outcome: Proportion of n-6 HUFA Arachidonic Acid (AA)
Description: as for outcome 5
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 6.25 (0.29) | 7.02 (0.22) | 6.37 (0.28)

7. Secondary Outcome: Proportion of n-6 HUFA Arachidonic Acid (AA)
Description: as for outcome 5
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 6.59 (0.30) | 7.27 (0.23) | 6.40 (0.28)

8. Secondary Outcome: Proportion of n-6 HUFA Arachidonic Acid (AA)
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 6.45 (0.29) | 7.02 (0.22) | 6.21 (0.28)

9. Secondary Outcome: Proportion of n-3 HUFA Eicosapentaenoic Acid (EPA)
Description: Tissue accretion of eicosapentaenoic acid (EPA or 20:5n3), an omega-3 (n-3) highly unsaturated fatty acid (HUFA), as measured in fasting plasma as a percent of total fatty acids.
Time Frame: Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 0.434 (0.065) | 0.455 (0.046) | 0.504 (0.062)

10. Secondary Outcome: Proportion of n-3 HUFA Eicosapentaenoic Acid (EPA)
Description: as for outcome 9
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 0.356 (0.061) | 0.479 (0.047) | 0.927 (0.061)

11. Secondary Outcome: Proportion of n-3 HUFA Eicosapentaenoic Acid (EPA)
Description: as for outcome 9
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 0.324 (0.064) | 0.452 (0.051) | 0.806 (0.061)

12. Secondary Outcome: Proportion of n-3 HUFA Eicosapentaenoic Acid (EPA)
Description: as for outcome 9
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 0.338 (0.061) | 0.388 (0.048) | 0.707 (0.062)

13. Secondary Outcome: Proportion of n-3 HUFA Docosahexaenoic Acid (DHA)
Description: Tissue accretion of Docosahexaenoic Acid (DHA or 22:6n3), an omega-3 (n-3) highly unsaturated fatty acid (HUFA), as measured in fasting plasma as a percent of total fatty acids.
Time Frame: Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 1.30 (0.11) | 1.16 (0.08) | 1.41 (0.11)

14. Secondary Outcome: Proportion of n-3 HUFA Docosahexaenoic Acid (DHA)
Description: as for outcome 13
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 1.39 (0.11) | 1.38 (0.08) | 2.25 (0.11)

15. Secondary Outcome: Proportion of n-3 HUFA Docosahexaenoic Acid (DHA)
Description: as for outcome 13
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 1.48 (0.11) | 1.44 (0.09) | 2.13 (0.11)

16. Secondary Outcome: Proportion of n-3 HUFA Docosahexaenoic Acid (DHA)
Description: as for outcome 13
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of total fatty acids
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
Number analyzed (Participants) | 16 | 28 | 17
Percentage of total fatty acids | 1.40 (0.11) | 1.38 (0.09) | 1.99 (0.11)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Diet A: Low Omega-3 (n-3) + High Linoleic Acid (LA) | Diet B: Low Omega-3 (n-3) + Low Linoleic Acid (LA) | Diet C: High Omega-3 (n-3) + Low Linoleic Acid (LA)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/29 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/29 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/29 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT01251887/Prot_SAP_000.pdf